CLINICAL TRIAL: NCT00051883
Title: Chemical Dependency and Smoking Cessation: Patient's Views
Brief Title: Chemical Dependency and Smoking Cessation: Patient's Views - 1
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Kimber Richter, PhD, University of Kansas Medical Center
Other Study IDs: NIDA-00450-1; K01-00450-1
Record Dates: First submitted 2003-01-17; First posted 2003-01-20 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to asses patient views on smoking cessation and tobacco harm reduction during drug treatment.

DETAILED DESCRIPTION:
Participants included 34 patients who had never voluntarily quit smoking for longer than 24 hours (continuous smokers), 34 smokers who had quit smoking for at least 24 hours before but had relapsed (relapsers), and 10 former smokers who had been abstinent for at least the past 6 months (successful quitters). We held 7 focus groups, 3 with continuous smokers and 4 with relapsers. Focus groups lasted 2 hours and were held at participants' clinics to preserve confidentiality. We conducted hour-long individual interviews with successful quitters. All participants completed a brief written survey immediately before their session. Survey items included questions on demographics, smoking behaviors, and motivation for cessation, reduction, and nicotine maintenance. We reimbursed all participants $40 and provided a meal to focus group attendees.

ELIGIBILITY:
Inclusion Criteria:

Selection criteria included being 18 years or older, smoking 5 or more cigarettes per day for at least 2 years, and being enrolled continuously in methadone maintenance treatment (MMT) for at least the past 2 years.

Exclusion Criteria:

Being less than 18 years of age, smoking 4 or fewer cigarettes per day, smoking less than daily for less than 2 years, and not being enrolled continuously in methadone treatment for at least the 2 past years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Substance abuse treatment patients
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 1999-12; Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimber Richter, Ph.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States